CLINICAL TRIAL: NCT01081678
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Determine the Efficacy, Safety, and Tolerability of AMG 785 in Adults With a Fresh Unilateral Hip Fracture, Status Post Surgical Fixation
Brief Title: Study To Assess FRacTure Healing With SclerosTin Antibody - Hip
Acronym: STARTT-Hip
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20080394
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Results first posted 2019-05-02 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Fracture Healing
Keywords: AMG 785; Proximal Femur; Fracture Healing; Hip Fracture
MeSH Terms: conditions — Hip Fractures | interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo to romosozumab administered by subcutaneous injection on day 1 and at weeks 2, 6, and 12.
  Interventions: Drug: Placebo
- Romosozumab 70 mg (Experimental): Participants received 70 mg romosozumab administered by subcutaneous injection on day 1 and at weeks 2, 6, and 12.
  Interventions: Drug: Romosozumab
- Romosozumab 140 mg (Experimental): Participants received 140 mg romosozumab administered by subcutaneous injection on day 1 and at weeks 2, 6, and 12.
  Interventions: Drug: Romosozumab
- Romosozumab 210 mg (Experimental): Participants received 210 mg romosozumab administered by subcutaneous injection on day 1 and at weeks 2, 6, and 12.
  Interventions: Drug: Romosozumab

INTERVENTIONS:
Drug: Placebo — Administered by subcutaneous (under the skin) injection
  Arms: Placebo
Drug: Romosozumab — Administered by subcutaneous injection
  Other Names: AMG 785; Evenity
  Arms: Romosozumab 140 mg; Romosozumab 210 mg; Romosozumab 70 mg

SUMMARY:
This is an international, multi-center study to determine the efficacy, safety, and tolerability of romosozumab (AMG 785) in adults with a fresh unilateral hip fracture, status post surgical fixation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 55 to 95 years
* fresh unilateral low energy intertrochanteric or femoral neck fracture as the primary injury, confirmed by X-ray and in the opinion of the treating surgeon amenable to repair by internal fixation
* internal fixation of the fracture with devices approved by local regulatory agency, performed no later than 7 days after injury for intertrochanteric or undisplaced femoral neck fractures and no later than 2 days after injury for displaced femoral neck fractures

  * intertrochanteric fracture: sliding hip screw or IM nail
  * femoral neck fracture: sliding hip screw or at least 3 cancellous screws

Exclusion Criteria:

* severe symptomatic osteoarthritis of the lower extremity
* inability to independently rise from armchair or walk 200 meters before hip fracture
* presence of concomitant injuries such as rib fractures, wrist fractures, or acute symptomatic vertebral fractures which severely impair the ability to rise from a chair
* associated extremity injuries including ipsilateral or contralateral fractures of the foot, tibia or fibula, wrist, humerus, femoral shaft, femoral head or hip dislocation, that may delay weight-bearing beyond one week after surgery
* head-injury, as defined by Glasgow Coma Scale < 13 prior to randomization
* use of bone grafts or bone substitutes at the time of fracture fixation
* major polytrauma or significant axial trauma, with Injury Severity Score > 16
* pathological fracture or history of metabolic or bone disease (except osteoporosis) that may interfere with the interpretation of the results, such as Paget's disease, rheumatoid arthritis, osteomalacia, osteopetrosis, ankylosing spondylitis, Cushing's disease, hyperprolactinemia
* history of symptomatic spinal stenosis that has not been surgically corrected. If surgically corrected, the subject must be asymptomatic to be eligible for the study.
* history of facial nerve paralysis
* malignancy (except fully resected cutaneous basal cell or squamous cell carcinoma, cervical carcinoma in situ) within the last 5 years
* history of solid organ or bone marrow transplants
* evidence of elevated transaminases (≥ 2.0 x upper limits of normal) or significantly impaired renal function (creatinine clearance of ≤ 30 mL/min)
* evidence of current hypercalcemia or hypocalcemia (outside of 1.1 x the normal range)
* bone morphogenic proteins (BMP)-2 or BMP-7 at the time of definitive fracture fixation

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2010-06-20 (Actual); Primary Completion 2012-06-30 (Actual); Study Completion 2013-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (92):
- United States (12):
  - Research Site, Birmingham, Alabama
  - Research Site, Pomona, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Indianapolis, Indiana
  - Research Site, Woodbury, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Brooklyn, New York
  - Research Site, Rochester, New York
  - Research Site, Altoona, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, State College, Pennsylvania
- Research Site, Buenos Aires, Argentina
- Australia (2):
  - Research Site, Liverpool, New South Wales
  - Research Site, Footscray, Victoria
- Belgium (5):
  - Research Site, Bruges
  - Research Site, Genk
  - Research Site, Leuven
  - Research Site, LiÃ¨ge
  - Research Site, Liège
- Bulgaria (3):
  - Research Site, Blagoevgrad
  - Research Site, Pleven
  - Research Site, Plovdiv
- Canada (8):
  - Research Site, Red Deer, Alberta
  - Research Site, Cambridge, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Denmark (4):
  - Research Site, Ã…rhus C
  - Research Site, Hvidovre
  - Research Site, KÃ¸benhavn NV
  - Research Site, Viborg
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (3):
  - Research Site, Kuopio
  - Research Site, Oulu
  - Research Site, Turku
- Germany (4):
  - Research Site, Aachen
  - Research Site, Berlin
  - Research Site, München
  - Research Site, Münster
- Greece (4):
  - Research Site, Athens
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szeged
- India (8):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Nashik, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
  - Research Site, Mangalore
  - Research Site, Nashik
- Italy (4):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Roma (RM)
  - Research Site, Verona
- Latvia (2):
  - Research Site, Riga
  - Research Site, Valmiera
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Haarlem
  - Research Site, Nieuwegein
- Research Site, Christchurch, New Zealand
- Poland (3):
  - Research Site, KrakÃ³w
  - Research Site, Lublin
  - Research Site, Warsaw
- Slovenia (4):
  - Research Site, Celje
  - Research Site, Izola
  - Research Site, Jesenice
  - Research Site, Šempeter pri Gorici
- Sweden (2):
  - Research Site, LinkÃ¶ping
  - Research Site, Lund
- Switzerland (4):
  - Research Site, Basel
  - Research Site, Lausanne
  - Research Site, Lucerne
  - Research Site, Zurich
- United Kingdom (5):
  - Research Site, Barnet
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Norwich

REFERENCES:
- [Background] Schemitsch EH, Miclau T, Karachalios T, Nowak LL, Sancheti P, Poolman RW, Caminis J, Daizadeh N, Dent-Acosta RE, Egbuna O, Chines A, Maddox J, Grauer A, Bhandari M. A Randomized, Placebo-Controlled Study of Romosozumab for the Treatment of Hip Fractures. J Bone Joint Surg Am. 2020 Apr 15;102(8):693-702. doi: 10.2106/JBJS.19.00790. PMID 31977817
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 63 centers in 22 countries in Eastern Europe, Western Europe, India, North America, Latin America, Australia, New Zealand and Hong Kong.
Pre-assignment Details: Participants were randomized in a 2:3:3:3 ratio to 1 of 3 romosozumab treatment groups or placebo.
  Randomization followed operative fracture repair and was stratified by type of fracture, type of fixation device and age at entry. There were 7 randomization strata.
Period: Overall Study
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Started | 89 | 60 | 93 | 90
Received Study Drug | 87 | 60 | 89 | 89
Completed 24 Weeks of Study | 73 | 50 | 72 | 68
Completed | 62 | 44 | 62 | 61
Not Completed | 27 | 16 | 31 | 29
Not completed — Ineligibility Determined | 0 | 0 | 1 | 1
Not completed — Noncompliance | 3 | 4 | 5 | 2
Not completed — Adverse Event | 2 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 15 | 7 | 17 | 14
Not completed — Administrative Decision | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 4 | 1 | 4 | 3
Not completed — Death | 2 | 2 | 2 | 6
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg | Total
Number analyzed (Participants) | 89 | 60 | 93 | 90 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.0 (8.6) | 76.6 (10.3) | 75.8 (10.1) | 76.7 (9.5) | 76.3 (9.5)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 10 | 8 | 17 | 11 | 46
  ≥ 65 years | 79 | 52 | 76 | 79 | 286
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 42 | 64 | 55 | 228
  Male | 22 | 18 | 29 | 35 | 104
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 77 | 52 | 81 | 70 | 280
  Black or African American | 0 | 0 | 0 | 1 | 1
  Hispanic or Latino | 0 | 1 | 1 | 0 | 2
  Asian | 12 | 7 | 11 | 19 | 49
Randomization Stratification [Count of Participants; unit: Participants] — Randomization was stratified by type of fracture (intertrochanteric vs. displaced femoral neck vs. undisplaced femoral neck), type of fixation device (sliding hip screw (SHS) vs. intramedullary (IM) nail vs. cancellous screws) and age at entry (55-75 years vs. ≥ 76 years).
  Participants
    Intertrochanteric, SHS and 55-75 years | 13 | 9 | 14 | 14 | 50
    Intertrochanteric, SHS and ≥ 76 years | 16 | 11 | 16 | 16 | 59
    Intertrochanteric, IM Nail and 55-75 years | 15 | 10 | 17 | 16 | 58
    Intertrochanteric, IM Nail and ≥ 76 years | 33 | 22 | 34 | 33 | 122
    Displaced femoral neck and SHS | 3 | 2 | 3 | 3 | 11
    Displaced femoral neck and cancellous screws | 6 | 4 | 6 | 5 | 21
    Undisplaced femoral neck | 3 | 2 | 3 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Timed-Up-and-Go (TUG) Over Week 6 Through Week 20
Description: Functional healing was measured by the timed-up-and-go test (TUG) over Weeks 6 through 20. During this assessment, the clinician timed the participant while they stood up from a seated position in a chair, walked three meters, turned around, walked three meters back to the chair, and returned to the seated position. A TUG value of ten seconds or less was considered normal for a healthy elderly person. Higher TUG values after hip fracture have been shown to be a predictor of future falls.
  Least squares mean (LSM) estimates were based on a repeated measures model fitted with the log-transformed TUG values at weeks 2, 6, 12, 16, 20, 24, 36, 52 as the dependent variable and adjusted for treatment, randomized strata, gender, country category, pre-fracture community-dwelling status, pre-fracture walking aid use, quality of surgical fixation, visit, and treatment-by-visit interaction and back-transformed using the exponential transformation.
Time Frame: Weeks 6, 12, 16, and 20
Population: Randomized participants who received at least one dose of study drug with available data at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 87 | 60 | 89 | 89
seconds
  Week 6: number analyzed (Participants) | 80 | 56 | 84 | 79
  Week 6 | 54.1 [44.4 to 66.0] | 41.0 [32.4 to 51.9] | 47.2 [38.9 to 57.4] | 53.3 [43.8 to 64.8]
  Week 12: number analyzed (Participants) | 75 | 53 | 82 | 75
  Week 12 | 29.8 [25.3 to 35.2] | 27.6 [22.7 to 33.5] | 30.0 [25.6 to 35.2] | 36.1 [30.7 to 42.5]
  Week 16: number analyzed (Participants) | 75 | 52 | 78 | 71
  Week 16 | 26.2 [22.2 to 30.8] | 23.3 [19.2 to 28.3] | 26.9 [23.0 to 31.6] | 31.8 [27.1 to 37.4]
  Week 20: number analyzed (Participants) | 75 | 52 | 75 | 70
  Week 20 | 23.8 [20.3 to 28.0] | 21.9 [18.1 to 26.6] | 22.9 [19.5 to 26.8] | 29.1 [24.8 to 34.2]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg vs Romosozumab 140 mg vs Romosozumab 210 mg; The primary analysis was based on a test for linear trend in dose response at weeks 6, 12, 16, and 20. To account for multiple comparisons over time points, the primary analysis used a size α = 0.05 F-test with 4 degrees of freedom for the contrasts at Weeks 6, 12, 16, and 20; Test type: Other; p = 0.1983, F-test; The p-value is based on F-test of multi-linear contrasts at Week 6 through Week 20

2. Secondary Outcome: Timed-Up-and-Go (TUG) at Each Visit
Description: During the timed-up-and-go test the clinician timed the participant while they stood up from a seated position in a chair, walked 3 meters, turned around, walked 3 meters back to the chair, and returned to a seated position. A TUG value of ≤ 10 seconds is considered normal for a healthy elderly person.
  LSMs were based on a repeated measures model adjusting for treatment, randomized strata, gender, country category, pre-fracture community-dwelling status, pre-fracture walking aid use, quality of surgical fixation, visit, and treatment-by-visit interaction.
  Missing TUG values for participants still on study were imputed using the last observation carried forward (LOCF) when possible. If no observation could be carried forward, the maximum TUG value observed among all participants at a given visit was used. TUG values obtained after unplanned revision surgery were replaced by carrying forward the last available observed or imputed value prior to unplanned revision surgery.
Time Frame: Weeks 2, 6, 12, 16, 20, 24, 36, and 52
Population: Randomized participants who received at least 1 dose of study drug. LOCF imputation was used when possible, as described above.
Measure: Least Squares Mean (95% Confidence Interval); unit: seconds
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 87 | 60 | 89 | 89
seconds
  Week 2: number analyzed (Participants) | 80 | 58 | 86 | 83
  Week 2 | 132.3 [111.0 to 153.6] | 119.3 [94.2 to 144.4] | 121.7 [101.0 to 142.5] | 129.8 [108.9 to 150.7]
  Week 6: number analyzed (Participants) | 80 | 56 | 84 | 79
  Week 6 | 92.4 [74.9 to 109.9] | 69.5 [48.6 to 90.4] | 80.3 [63.1 to 97.5] | 86.7 [69.3 to 104.0]
  Week 12: number analyzed (Participants) | 75 | 53 | 82 | 75
  Week 12 | 47.4 [37.6 to 57.1] | 39.1 [27.4 to 50.7] | 44.6 [35.1 to 54.1] | 56.3 [46.6 to 65.9]
  Week 16: number analyzed (Participants) | 75 | 52 | 78 | 71
  Week 16 | 43.1 [34.1 to 52.1] | 31.6 [20.9 to 42.4] | 39.7 [30.9 to 48.6] | 50.1 [41.2 to 59.1]
  Week 20: number analyzed (Participants) | 75 | 52 | 75 | 70
  Week 20 | 36.4 [28.3 to 44.6] | 31.0 [21.2 to 40.7] | 35.1 [27.1 to 43.1] | 45.6 [37.5 to 53.8]
  Week 24: number analyzed (Participants) | 73 | 51 | 73 | 68
  Week 24 | 33.3 [25.8 to 40.7] | 28.9 [20.1 to 37.8] | 31.7 [24.4 to 39.0] | 40.9 [33.5 to 48.4]
  Week 36: number analyzed (Participants) | 71 | 50 | 68 | 66
  Week 36 | 32.4 [25.1 to 39.7] | 26.3 [17.5 to 35.0] | 29.8 [22.5 to 37.0] | 38.7 [31.3 to 46.0]
  Week 52: number analyzed (Participants) | 66 | 48 | 67 | 63
  Week 52 | 28.7 [22.2 to 35.1] | 22.8 [15.2 to 30.5] | 28.8 [22.5 to 35.2] | 36.3 [29.8 to 42.7]

3. Secondary Outcome: Time to Radiographic Healing
Description: Time to radiographic healing is the time interval from the surgery date for the eligible hip fracture to the date of radiographic healing, defined as effacement of the fracture lines by newly formed bone along the cortices and within the trabecular bone on anteroposterior and lateral (or oblique) radiographs. Radiographic fracture healing was determined by a panel of independent reviewers blinded to treatment.
  The cumulative incidence function (CIF) method was used to estimate the median time to radiographic healing and the confidence intervals. Unplanned revision surgery to promote healing was considered a competing risk in CIF estimate.
Time Frame: 52 weeks
Population: All randomized participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 87 | 60 | 89 | 89
weeks | 16.4 [15.3 to 20.1] | 16.9 [12.9 to 20.3] | 16.6 [13.3 to 17.1] | 16.9 [13.3 to 20.9]

4. Secondary Outcome: Radiographic Union Scale for Hip (RUSH) Score At Each Visit
Description: The radiographic Union Scale for Hip (RUSH) is a semiquantitative scoring assessment to assess hip fracture healing after surgical repair. The RUSH has 4 key domains based on radiographic parameters used by orthopedic surgeons and radiologists in routine clinical practice including cortical bridging (4 to 12 points), cortical fracture line disappearance (4 to 12 points), trabecular consolidation (1 to 3 points), and trabecular index disappearance of fracture line (1 to 3 points). The score has a minimum of 10 points (definitely not healed) and a maximum of 30 points (definitely healed).
Time Frame: Weeks 2, 6, 12, 16, 20, 24, 36, and 52
Population: Randomized participants who received at least 1 dose of study drug, with available data at baseline and at each time point. Missing RUSH scores for participants who were still on study were imputed using the using last observation carried forward procedure when possible.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 87 | 60 | 89 | 89
units on a scale
  Week 2: number analyzed (Participants) | 76 | 51 | 78 | 75
  Week 2 | 12.1 (3.3) | 12.7 (3.5) | 12.1 (3.4) | 12.0 (3.1)
  Week 6: number analyzed (Participants) | 79 | 55 | 81 | 78
  Week 6 | 18.1 (3.6) | 18.0 (4.2) | 18.4 (3.4) | 18.3 (4.0)
  Week 12: number analyzed (Participants) | 74 | 53 | 80 | 74
  Week 12 | 23.3 (4.6) | 22.8 (4.8) | 22.9 (4.8) | 22.3 (5.3)
  Week 16: number analyzed (Participants) | 74 | 52 | 77 | 69
  Week 16 | 25.6 (4.3) | 25.7 (4.5) | 25.5 (5.0) | 25.5 (4.7)
  Week 20: number analyzed (Participants) | 75 | 52 | 74 | 68
  Week 20 | 26.8 (4.1) | 27.3 (4.1) | 27.4 (4.0) | 26.4 (4.6)
  Week 24: number analyzed (Participants) | 73 | 51 | 73 | 67
  Week 24 | 27.8 (3.4) | 27.8 (3.9) | 28.3 (3.5) | 27.3 (3.9)
  Week 36: number analyzed (Participants) | 71 | 50 | 67 | 65
  Week 36 | 28.7 (2.6) | 28.3 (3.6) | 29.1 (2.1) | 28.2 (3.5)
  Week 52: number analyzed (Participants) | 65 | 48 | 66 | 62
  Week 52 | 29.4 (2.0) | 28.5 (3.8) | 29.6 (1.8) | 28.7 (3.3)

5. Secondary Outcome: Harris Hip Score At Each Visit
Description: The Harris Hip Score is a clinician-based outcome that assesses pain, function, deformity, and range of motion. The pain domain measures pain severity and its effect on activities and need for pain medication. The function domain consists of daily activities and gait. Deformity takes into account hip flexion, adduction, internal rotation, and extremity length discrepancy. Range of motion measures hip flexion, abduction, external and internal rotation, and adduction. The score ranges form 0-100 (best possible outcome) covering pain (0-44 points), function (0-47 points), absence of deformity (4 points), and range of motion (5 points). LSMs were based on a repeated measures model fitted with the Harris hip score values at weeks 2, 6, 12, 16, 20, 24, 36, and 52 as the dependent variable and adjusted for treatment, randomized strata, gender, pre-fracture community-dwelling status, pre-fracture walking aid use, quality of surgical fixation, visit, and treatment-by-visit interaction.
Time Frame: Weeks 2, 6, 12, 16, 20, 24, 36, and 52
Population: Randomized participants who received at least 1 dose of study drug with available data at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 87 | 60 | 89 | 89
units on a scale
  Week 2: number analyzed (Participants) | 77 | 56 | 82 | 79
  Week 2 | 46.6 [43.1 to 50.1] | 47.7 [43.6 to 51.9] | 47.3 [43.9 to 50.8] | 46.5 [43.1 to 50.0]
  Week 6: number analyzed (Participants) | 76 | 53 | 78 | 71
  Week 6 | 58.6 [55.1 to 62.1] | 62.5 [58.3 to 66.7] | 61.6 [58.1 to 65.0] | 59.5 [55.9 to 63.0]
  Week 12: number analyzed (Participants) | 73 | 51 | 68 | 68
  Week 12 | 71.2 [67.9 to 74.5] | 70.9 [67.0 to 74.9] | 71.7 [68.3 to 75.1] | 69.6 [66.2 to 72.9]
  Week 16: number analyzed (Participants) | 68 | 48 | 71 | 64
  Week 16 | 74.1 [70.8 to 77.4] | 76.5 [72.6 to 80.5] | 76.1 [72.7 to 79.4] | 72.8 [69.4 to 76.2]
  Week 20: number analyzed (Participants) | 64 | 43 | 69 | 62
  Week 20 | 76.2 [73.0 to 79.3] | 80.2 [76.4 to 83.9] | 80.5 [77.4 to 83.6] | 77.5 [74.3 to 80.7]
  Week 24: number analyzed (Participants) | 66 | 42 | 62 | 59
  Week 24 | 79.0 [76.2 to 81.8] | 80.3 [76.8 to 83.7] | 83.0 [80.1 to 85.8] | 80.1 [77.2 to 83.0]
  Week 36: number analyzed (Participants) | 62 | 45 | 60 | 60
  Week 36 | 80.3 [77.0 to 83.6] | 82.0 [78.1 to 85.8] | 86.8 [83.5 to 90.2] | 83.6 [80.2 to 86.9]
  Week 52: number analyzed (Participants) | 59 | 41 | 60 | 58
  Week 52 | 84.3 [81.3 to 87.4] | 86.7 [83.0 to 90.3] | 89.0 [85.9 to 92.1] | 83.8 [80.7 to 86.9]

6. Secondary Outcome: Hip Pain Score at Each Visit
Description: Hip pain was assessed using a visual analog scale (VAS). Participants were asked to rate their pain as a result of the hip fracture on a 100 mm vertical scale with 0 indicating no pain at all and 100 indicating the worst pain they could imagine.
  LSMs were based on a repeated measures model fitted with hip pain score values at weeks 2, 6, 12, 16, 20, 24, 36, and 52 as the dependent variable and adjusted for treatment, randomized strata, gender, pre-fracture community-dwelling status, pre-fracture walking aid use, quality of surgical fixation, visit, and treatment-by-visit interaction.
Time Frame: Weeks 2, 6, 12, 16, 20, 24, 36, and 52
Population: Randomized participants who received at least 1 dose of study drug with available data at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Number analyzed (Participants) | 87 | 60 | 89 | 89
units on a scale
  Week 2: number analyzed (Participants) | 74 | 53 | 80 | 77
  Week 2 | 34.3 [28.2 to 40.4] | 33.1 [25.9 to 40.3] | 40.3 [34.4 to 46.2] | 43.0 [37.1 to 48.9]
  Week 6: number analyzed (Participants) | 73 | 51 | 76 | 71
  Week 6 | 26.3 [20.8 to 31.7] | 19.5 [13.1 to 26.0] | 25.1 [19.7 to 30.4] | 27.5 [22.1 to 32.9]
  Week 12: number analyzed (Participants) | 70 | 50 | 67 | 68
  Week 12 | 19.4 [14.1 to 24.8] | 17.8 [11.5 to 24.1] | 17.5 [12.1 to 22.8] | 23.7 [18.3 to 29.0]
  Week 16: number analyzed (Participants) | 67 | 46 | 71 | 64
  Week 16 | 18.1 [13.0 to 23.3] | 13.5 [7.4 to 19.6] | 16.8 [11.8 to 21.8] | 17.4 [12.2 to 22.5]
  Week 20: number analyzed (Participants) | 62 | 43 | 68 | 62
  Week 20 | 15.8 [11.2 to 20.4] | 9.2 [3.8 to 14.7] | 14.0 [9.5 to 18.5] | 15.0 [10.5 to 19.6]
  Week 24: number analyzed (Participants) | 65 | 42 | 61 | 59
  Week 24 | 13.8 [9.6 to 18.0] | 9.1 [4.0 to 14.2] | 12.7 [8.4 to 17.0] | 13.1 [8.8 to 17.3]
  Week 36: number analyzed (Participants) | 62 | 45 | 60 | 60
  Week 36 | 14.3 [9.6 to 19.0] | 10.9 [5.4 to 16.4] | 11.6 [6.8 to 16.3] | 10.2 [5.5 to 14.9]
  Week 52: number analyzed (Participants) | 59 | 40 | 61 | 58
  Week 52 | 13.4 [9.2 to 17.7] | 7.2 [2.1 to 12.3] | 9.3 [5.1 to 13.5] | 10.4 [6.2 to 14.6]

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Romosozumab 70 mg | Romosozumab 140 mg | Romosozumab 210 mg
Serious Adverse Events (participants affected / at risk) | 25/87 | 9/60 | 15/89 | 26/89
Other Adverse Events (participants affected / at risk) | 31/87 | 24/60 | 30/89 | 26/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | Romosozumab 70 mg (N=60) | Romosozumab 140 mg (N=89) | Romosozumab 210 mg (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 1 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Haemorrhage coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 0 | 1 | 0
Device failure (General disorders) | 0 | 0 | 0 | 1
Medical device complication (General disorders) | 0 | 1 | 0 | 1
Medical device discomfort (General disorders) | 0 | 1 | 0 | 0
Medical device pain (General disorders) | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 3 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 3
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cerebellar artery thrombosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1
Dementia Alzheimer's type (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Nail operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=87) | Romosozumab 70 mg (N=60) | Romosozumab 140 mg (N=89) | Romosozumab 210 mg (N=89)
Constipation (Gastrointestinal disorders) | 11 | 6 | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 2 | 2 | 4
Nausea (Gastrointestinal disorders) | 7 | 4 | 7 | 2
Pyrexia (General disorders) | 0 | 3 | 2 | 3
Urinary tract infection (Infections and infestations) | 8 | 4 | 8 | 4
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 5 | 1 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3 | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 7 | 5 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 2
Hypertension (Vascular disorders) | 3 | 4 | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.